CLINICAL TRIAL: NCT00522028
Title: Asymptomatic Primary Hyperparathyroidism: A Prospective, Randomized Trial
Acronym: SIPH
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Rikshospitalet University Hospital (Other); Göteborg University (Other); Rigshospitalet, Denmark (Other); Karolinska University Hospital (Other); Uppsala University Hospital (Other); Haukeland University Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Jens Bollerslev, Professor, Oslo University Hospital
Other Study IDs: S-96107 (REK); 9571 (NSD) (Other: Oslo University Hospital)
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 1996-06

CONDITIONS: Primary Hyperparathyroidism
Keywords: QoL; Osteodensitometry; Arterial pressure; PTH
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study is a randomized, controlled trial that investigates the effects of parathyroidectomy or medical observation in mild asymptomatic pHPT on morbidity and quality of life (QoL).

DETAILED DESCRIPTION:
The patients are included and randomized by block randomization to medical observation or parathyroidectomy by an experienced parathyroid surgeon.

The patients will be followed up for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, asymptomatic pHPT
* 2.60>S-Ca<2.85 mmol/liter
* Age between 50 and 80 yr
* No medications interfering with Ca-metabolism
* Informed consent

Exclusion Criteria:

* Hyperparathyroid bone disease
* Previous operation in the neck
* Impaired kidney function
* Kidney stones
* Complicating medical conditions
* Psychiatric disorders
* Multiple endocrine neoplasia,
* Familial hypocalcuric hypercalcemia
* Familial HPT

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 1998-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bollerslev, MD, Principal Investigator — Rikshospitalet University Hospital
Locations (1):
- Oslo University Hospital - Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Result] Bollerslev J, Jansson S, Mollerup CL, Nordenstrom J, Lundgren E, Torring O, Varhaug JE, Baranowski M, Aanderud S, Franco C, Freyschuss B, Isaksen GA, Ueland T, Rosen T. Medical observation, compared with parathyroidectomy, for asymptomatic primary hyperparathyroidism: a prospective, randomized trial. J Clin Endocrinol Metab. 2007 May;92(5):1687-92. doi: 10.1210/jc.2006-1836. Epub 2007 Feb 6. PMID 17284629
- [Result] Bollerslev J, Rosen T, Mollerup CL, Nordenstrom J, Baranowski M, Franco C, Pernow Y, Isaksen GA, Godang K, Ueland T, Jansson S; SIPH Study Group. Effect of surgery on cardiovascular risk factors in mild primary hyperparathyroidism. J Clin Endocrinol Metab. 2009 Jul;94(7):2255-61. doi: 10.1210/jc.2008-2742. Epub 2009 Apr 7. PMID 19351725
- [Result] Persson A, Bollerslev J, Rosen T, Mollerup CL, Franco C, Isaksen GA, Ueland T, Jansson S, Caidahl K; SIPH Study Group. Effect of surgery on cardiac structure and function in mild primary hyperparathyroidism. Clin Endocrinol (Oxf). 2011 Feb;74(2):174-80. doi: 10.1111/j.1365-2265.2010.03909.x. PMID 21044114
- [Result] Lundstam K, Heck A, Mollerup C, Godang K, Baranowski M, Pernow Y, Varhaug JE, Hessman O, Rosen T, Nordenstrom J, Jansson S, Hellstrom M, Bollerslev J; SIPH Study Group. Effects of parathyroidectomy versus observation on the development of vertebral fractures in mild primary hyperparathyroidism. J Clin Endocrinol Metab. 2015 Apr;100(4):1359-67. doi: 10.1210/jc.2014-3441. Epub 2015 Jan 30. PMID 25636048
- [Derived] Heck A, Pretorius M, Lundstam K, Godang K, Hellstrom M, Ueland T, Bollerslev J. No effect of surgery on kidney and cardiovascular risk factors in mild primary hyperparathyroidism: secondary analyses from a 10-year randomized controlled trial. Eur J Endocrinol. 2024 Aug 30;191(3):354-360. doi: 10.1093/ejendo/lvae109. PMID 39189547
- [Derived] Pretorius M, Lundstam K, Heck A, Fagerland MW, Godang K, Mollerup C, Fougner SL, Pernow Y, Aas T, Hessman O, Rosen T, Nordenstrom J, Jansson S, Hellstrom M, Bollerslev J. Mortality and Morbidity in Mild Primary Hyperparathyroidism: Results From a 10-Year Prospective Randomized Controlled Trial of Parathyroidectomy Versus Observation. Ann Intern Med. 2022 Jun;175(6):812-819. doi: 10.7326/M21-4416. Epub 2022 Apr 19. PMID 35436153